CLINICAL TRIAL: NCT00494962
Title: An Open-Label, Single-Dose, Randomized, 2-Period, Crossover, Bioequivalence Study Between Two 5-mg Tablets and a New 10-mg Tablet Formulation of Lecozotan SR in Healthy Subjects.
Brief Title: Study Comparing Lecozotan SR Two 5-mg Tablets Vs. Lecozotan SR One 10-mg Tablet in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 3098B1-1147
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan

INTERVENTIONS:
Drug: lecozotan SR

SUMMARY:
To determine the bioequivalence between two 5-mg tablets of lecozotan and the new 10-mg tablet of lecozotan.

ELIGIBILITY:
Inclusion criteria:

* Generally healthy, man and women, aged 18 to 50 years.

Exclusion criteria:

* History or active presence of clinically important medical disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2007-06; Study Completion 2007-06

PRIMARY OUTCOMES:
Pharmacokinetic (PK) analyses

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com
Locations (1):
- Neuss, Germany